CLINICAL TRIAL: NCT01761721
Title: Robot-assisted Laparoscopic Hysterectomy-RALH- Postoperative Complications, Quality of Life and Health Economics
Acronym: RALH
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: H-2-2012-FSP26
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Endometrial Cancer; Treatment by Robotic Assisted Laparoscopy Hysterectomy
Keywords: Endometrial cancer (MeSH); Robotics (MeSH)
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RAHL: Women suspected of endometrial cancer planned to be treated by robotic assisted laparoscopy hysterectomy

SUMMARY:
The propose of this study is to describe recovery and experience of pain and health related quality of life after robot-assisted laparoscopic hysterectomy for women with Endometrial Cancer or Atypical Complex Hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

Women suspected of having Endometrial Cancer or having Atypical Complex hyperplasia

* Ability to understand and speak Danish
* Ability to cooperate
* Provision of written informed consent

Exclusion Criteria:

* Having a benign condition after histopathology postoperatively
* Bing assigned to radiation or chemotherapy postoperatively

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women suspected of endometrial cancer and treated with robot-assisted laparoscopic hysterectomy at Copenhagen University Hospital, Herlev.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2013-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Postoperative complications Postoperative complications Postoperative complications Postoperative complications | 0-4 months follow-up
  Postoperative complications demanding treatment

SECONDARY OUTCOMES:
Postoperative pain | 0-4 months follow-up
  Postoperative pain measured by Brief Pain Inventory, baseline, 1 and 5 weeks and 4 months postoperatively
Health Related Quality of Life | 0-4 months follow-up
  Health Related Quality of Life measured by QlQ-C30 and EN 24 (EORTC), EQ -5D, baseline, 1 and 5 weeks and 4 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne F Herling, RN; MHSc, Principal Investigator — Department of Anaesthesiology, Copenhagen University Hospital, Herlev
Locations (1):
- Department of Anaesthesiology, Copenhagen University Hospital, Herlev, Herlev, Herlev, Denmark

REFERENCES:
- [Result] Herling SF, Moller AM, Palle C, Thomsen T. Health-related quality of life after robotic-assisted laparoscopic hysterectomy for women with endometrial cancer--A prospective cohort study. Gynecol Oncol. 2016 Jan;140(1):107-13. doi: 10.1016/j.ygyno.2015.10.024. Epub 2015 Nov 2. PMID 26541978